CLINICAL TRIAL: NCT01308359
Title: Impact of Glucose Administration on Perception of Fetal Movements
Brief Title: Use of Glucose and Saline for Fetal Movement Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Ariel Many, MD, Dep. of OB&GYN, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-10-am-0512-CTIL
Record Dates: First submitted 2010-12-14; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Fetal Movement Perception
Keywords: fetal movement
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- glucose 5% (Experimental): glucose 5%
  Interventions: Drug: IV glucose 5%
- saline (Active Comparator): saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: IV glucose 5% — 500 ml glucose 5% within 30 minutes
  Arms: glucose 5%
Drug: saline — saline
  Arms: saline

SUMMARY:
The purpose of this study is to investigate the hypothesis that glucose administration increases fetal movement perception by the pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients with singleton pregnancy during 3rd trimester

Exclusion Criteria:

* Any maternal medical condition (Diabetes, hypertension), multiple pregnancy, fetal anomaly, polyhydramnios

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
fetal movements as perceived by the mother | one hour
  Effect of glucose versus saline infusion on the perception of fetal movements. the mother will count fetal movements that she feels one hour following saline/glucose infusion and report to the obstetrician in charge. The research aims to clarify whether glucose increases fetal movements.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Many, MD, Principal Investigator — Lis Maternity Hospital
Locations (1):
- Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel